CLINICAL TRIAL: NCT05499091
Title: Functional Study to Indentify Genetic Etiology of Rare Diseases - ORIGIN
Acronym: ORIGIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 49RC22_0061
Record Dates: First submitted 2022-07-13; First posted 2022-08-12 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Rare Diseases; Genetic Disease
MeSH Terms: conditions — Rare Diseases; Genetic Diseases, Inborn | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: In addition to the standard clinical care, blood samples and/or urine samples and/or skin biopsy will be proposed to the included patient to carry out further genetic analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study Arm (Experimental): Specific interventions:
  Blood samples, skin biopsy, urine collection or operational waste qualified as research sample.
  Interventions: Procedure: Skin biopsy, blood sample, urine sample

INTERVENTIONS:
Procedure: Skin biopsy, blood sample, urine sample — blood samples, urine samples, skin samples.

SUMMARY:
Next generation sequencing (NGS) allows some better diagnostic results, particularly, in the rare diseases field. At a twenty five percent rate, those exams highlight some variants which are not yet described in human pathology. The relationship between a variant found inside a candidate gene and a pathology, is able to be confirmed by functional studies at a protein level. This study aims to build a biological collection to feed further functional studies to confirm the relationship between NGS identified variants, and the clinical signs and symptoms.

ELIGIBILITY:
Inclusion Criteria:

Patient :

* Child or adult affected by a rare disease whose molecular functions are not known, or whose pathophysiologic mechanism are not fully understood.
* Patient included inside the BaMaRa (French rare disease national data bank) database dedicated to the rare diseases.
* Patient Affiliated to the French social security system.
* Patient consent form or legal representative consent form obtained.

Patient's parent :

* Parent of a patient affected by a rare disease whose molecular functions are not known, or whose pathophysiologic mechanism are not fully understood.
* Parent included in the BaMaRa database.
* Parent affiliated to the French social security system.
* Parent consent form obtained for himself/herself.

Patient's brother or sister :

* Brother or sister of a patient (underage or adult) affected by a rare disease whose molecular functions are not known, or whose pathophysiologic mechanism are not fully understood.
* Brother or sister included in the BaMaRa database.
* Brother or sister affiliated to the French social security system.
* Brother or sister consent form obtained for themselves or from their legal representative.

Exclusion Criteria:

* Poor understanding of the French language
* Legal of administrative liberty deprivation
* Psychiatric force care

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2042-10-10 (Estimated); Study Completion 2045-10-10 (Estimated)

PRIMARY OUTCOMES:
Identification of at least 80 new genes implicated in rare diseases via high-throughput sequencing technics and through functional studies. | 23 years
  Candidate genes, suspected to be responsible for rare diseases will be identified before the inclusion, during standard medical care, by exome or genome sequencing.
Collecting biological samples to build up a biobank | 23 years
  After a candidat gene identification, patient will be proposed sampling (blood or urine) or if a skin biopsy, an amniotic fluid puncture or any surgery are done during standard care, the remaing tissue or fluid, or operative wastes will be eligible too, to be stored in the biobank.
Candidat gene validation through functional studies. | 23 years
  Biological samples from the biobank will be made available after the study, to some specialized research teams, in order to validate or overturn those previously gene candidates by the way of some biological technics.

CONTACTS AND LOCATIONS:
Overall Officials: Estelle COLIN, MD-PhD, Principal Investigator — escolin@chu-angers.fr
Locations (1):
- Centre Hospitalo-Universitaire d'Angers, Angers, France

IPD SHARING:
Plan to Share IPD: Undecided